CLINICAL TRIAL: NCT05759650
Title: Validation of an Integrated Assessment Protocol for the Analysis of Functional Performance in Subjects With Obesity During Motor Tasks Associated With Daily and Work Activities. Pilot Study
Brief Title: Analysis of Functional Performance in Subjects With Obesity During Motor Tasks.
Acronym: Obesity_TASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 31C211
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analyses of Kinematic and Kinetic parameters of movement (Experimental)
  Interventions: Other: Execution of different motor tasks typical of daily life and work

INTERVENTIONS:
Other: Execution of different motor tasks typical of daily life and work — Patients with obesity will carry out different motor tasks typical of daily life and work and, using optoelectronic systems based on passive markers, force platforms and electromyographic systems, kinematic and kinetic parameters of movement will be recorded and analysed for the implementation of an integrated protocol for the clinical evaluation of subjects with obesity.

SUMMARY:
Background. Individuals with obesity can present several functional limitations that can significantly impact on their quality of life. Furthermore, even during the execution of specific motor tasks, subjects with obesity can experience excessive biomechanical overload. It is therefore necessary to develop appropriate assessment protocols that are able to provide support for risk assessment, in consideration of different types of motor tasks, including movements that can reflect the main daily and / or work activities. In this perspective, it is essential to define a protocol that includes an integrated evaluation process based on objective and quantitative metrics, i.e., functional scales, clinical scores, etc. In this context, the quantitative analysis of movement is widely used in clinical practice and in research to investigate in an objective and comprehensive way on movement disorders in various pathological conditions, including obesity. Conventionally, kinematic and kinetic parameters of movement are measured in motion analysis laboratories, using optoelectronic systems based on passive markers, force platforms and electromyographic systems, which represent the gold standard. Although motion analysis is considered accurate, the availability of specific laboratories, high costs and dependence on trained users sometimes limit its use in clinical practice. A variety of wearable sensors available today has enabled researchers and clinicians to pursue applications where individuals are monitored in home and outpatient settings.

Hypothesis and significance. The hypothesis is that wearables could reveal a good agreement, accuracy, and correlation between the parameters measured by means of optoelectronic system and those measured by wearables in individuals with obesity.

Specific Aims. The main objective is the implementation of an integrated protocol for the clinical evaluation of subjects with obesity through the analysis of the execution of different motor tasks typical of daily life and work. Appropriately identified clinical scores and scales will also be supported by quantitative evaluations carried out with human movement analysis systems (optoelectronic systems based on markers and inertial measurement units).

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 30/35 Kg/m2;
* No impediments to physical activity;

Exclusion Criteria:

* Pathologies of the locomotor system,
* Neurological pathologies affecting movement;
* Internal pathologies contraindicating physical activity;
* Pregnant or breastfeeding women;
* Individuals with genetic obesity (Down's or Prader-Willi syndrome).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Baseline balance and functional mobility | same day of intervention
  Measurement of balance and functional mobility using Timed Up and Go test (TUG) at baseline.

SECONDARY OUTCOMES:
Joint kinematics data aquisition | same day of intervention
  Joint kinematics data deriving from the use of optoelectronic systems and inertial measurement units will be collected, including trunk angles during flexion movement, axial rotation bending, upper limb flexion angle during lateral lift and angle on the frontal plane of the upper limb during front lift.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Cimolin, PhD, Study Director — Politecnico di Milano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Oggebbio, VB, Italy